CLINICAL TRIAL: NCT06970262
Title: FMT for Lung and Associated-organ Rescue Efficacy in Pulmonary Infection With MDROs: A Single-Center, Open-Label, Randomized Controlled Trial
Brief Title: FMT for Lung and Associated-organ Rescue Efficacy in Pulmonary Infection With MDROs
Acronym: FLARE-PM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jiancheng Zhang, Prof. Jiancheng Zhang, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0928-01
Record Dates: First submitted 2025-04-24; First posted 2025-05-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Lung Infection; Microbial Colonization; Food Intolerance Syndromes
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT intervention group (Experimental): On the basis of the standard ICU treatment protocol, FMT was administered via a nasojejunal tube. Over three consecutive days, 50-100 ml of intestinal flora suspension was delivered through the nasojejunal tube daily between 11:00 and 13:00.
  A strict antibiotic intervention window spans 24 hours before to 48 hours after FMT infusion. During this period, narrow-spectrum antibiotics active against confirmed pulmonary target MDROs (based on susceptibility testing) may continue to ensure effective infection control and patient safety. All broad-spectrum antibiotics should be stopped unless they are the only effective option. Empiric or prophylactic antibiotics without confirmed infection are prohibited. Oral vancomycin, metronidazole, and microbiota-disrupting quinolones should be avoided, except when intravenous quinolones are required for MDRO treatment. Antifungals may continue due to minimal impact on gut bacteria.
  Interventions: Other: Fecal suspension
- Control group (No Intervention): Receiving the standard ICU treatment protocol involves a comprehensive set of systematic and standardized medical and nursing interventions designed for critically ill patients in the ICU. These interventions are aimed at ensuring patient stability through multidisciplinary collaboration, continuous physiological monitoring, and functional support, while also facilitating recovery. The ICU treatment protocol is developed based on modern medical principles and extensive clinical experience, encompassing all aspects from fundamental care to advanced life support.
  The control group follows the same antibiotic rules during the same window but receives placebo. This ensures comparable anti-infective treatment intensity between groups.

INTERVENTIONS:
Other: Fecal suspension — Prepare 300 ml of intestinal flora suspension from 100-150 g of feces. Subjects can eat and drink freely during preparation but must fast for at least 2 hours before FMT (water allowed). No food or water is permitted within 2 hours after FMT.
  Arms: FMT intervention group

SUMMARY:
Currently, lung infections caused by multidrug-resistant organisms (MDROs) represent a significant global health burden. In the intensive care unit (ICU), the administration of antibiotics, opioids, proton pump inhibitors (PPIs), vasoconstrictors, and parenteral nutrition-combined with the underlying severity of critical illness-leads to profound disruption of the gut microbiota, which may concurrently impair pulmonary microecology and negatively influence long-term patient outcomes. Although pulmonary microecology has garnered increasing scientific attention, the potential causal link between gut dysbiosis and the development of pulmonary microbial imbalance remains poorly elucidated. As such, it is currently unclear whether gut dysbiosis in patients with MDRO-related pulmonary infection contributes to or exacerbates pulmonary microecological disturbances. This study aims to characterize differences in gut microbiota composition and pulmonary microecology between ICU patients with and without MDRO-associated pulmonary infection, and to investigate the association between alterations in gut microbiota and changes in the pulmonary microbial environment.

Fecal microbiota transplantation (FMT) is a therapeutic intervention involving the transfer of functionally intact microbial communities from healthy donors to recipients, with the objective of restoring a disrupted gut microbiota and treating both gastrointestinal and systemic conditions. Evidence suggests that FMT effectively reduces intestinal colonization by MDROs and prevents secondary infections in non-ICU populations. Over the past decade, FMT has demonstrated transformative potential in managing refractory intestinal and extra-intestinal diseases, offering a novel, mechanism-driven strategy for modulating host microbial ecosystems. These findings indicate that FMT not only facilitates the restoration of a balanced gut microbiota but may also reduce recurrent infections by suppressing the proliferation of drug-resistant bacterial strains. Given that gut-resident microorganisms serve as a major reservoir for enterogenic infections, hospital-acquired bacteremia, and ventilator-associated pneumonia, this project will conduct a prospective, randomized controlled trial (RCT) in critically ill patients admitted to the ICU with pulmonary infection-specifically targeting those eligible for antibiotic de-escalation and exhibiting clinical features of food intolerance syndrome. FMT will be administered via a nasojejunal tube to correct gut dysbiosis induced by broad-spectrum antimicrobials and other iatrogenic factors. The primary objectives are to evaluate the efficacy and safety of FMT in promoting the restoration of pulmonary microbial homeostasis and to assess its impact on clinically relevant outcomes, including length of stay in the ICU, ICU mortality, in-hospital mortality, and 28-day all-cause mortality.

ELIGIBILITY:
The initial step involves characterizing alterations in the pulmonary and intestinal microbiota among ICU patients with pathogen-associated infections, including multidrug-resistant organisms (MDROs), and examining the associations between these microbial changes.

Inclusion Criteria:

1. Age ranging from 18 to 70 years old;
2. Gender and ethnicity are not restricted;
3. Informed consent obtained.

Exclusion Criteria:

1. Airway antibiotics (administered via nebulization or intravenous infusion) have been utilized since the current hospitalization;
2. Pulmonary infection caused by non-bacterial pathogens, such as viruses, fungi, or atypical organisms;
3. Infections located outside the pulmonary system, including those in the bloodstream, abdominal cavity, or urinary tract;
4. Respiratory failure secondary to non-pulmonary infections, such as cardiogenic factors or sepsis-like syndromes;
5. Chronic pulmonary conditions, including chronic obstructive pulmonary disease (COPD), asthma, bronchiectasis, and pulmonary interstitial fibrosis;
6. Chronic gastrointestinal disorders, such as inflammatory bowel disease (IBD), irritable bowel syndrome (IBS), celiac disease, and non-alcoholic fatty liver disease (NAFLD);
7. Recent surgical procedures involving the abdomen or lungs (within 14 days prior to admission);
8. Pregnant or lactating individuals；
9. Subjects who participated in other clinical studies as trial participants at the time of enrollment or within 3 months prior to enrollment；
10. Lack of a signed written informed consent form.

Further trial will be conducted to investigate the effect and safety of FMT on the recovery of pulmonary microecological imbalance in critically ill patients, and to evaluate its impact on the length of stay in the ICU, ICU mortality, in-hospital mortality, and 28-day mortality, etc.

Inclusion Criteria:

1. Age 18-70 years, regardless of gender or ethnicity;
2. ICU admission ≥24 hours;
3. Expected ICU stay ≥7 days;
4. Mechanically ventilated patients with confirmed pulmonary MDRO infection prior to enrollment. Target MDRO has available narrow-spectrum antibiotics; if the pathogen is pan-resistant (e.g., pan-drug-resistant Acinetobacter baumannii) and treatment relies solely on polymyxins or other limited options, exclusion is required. The attending physician must confirm that short-term discontinuation of broad-spectrum antibiotics is safe;
5. Written informed consent provided.

Exclusion Criteria:

1. Severe systemic infection during early resuscitation, with hemodynamic instability, severe tissue hypoperfusion, or major electrolyte and acid-base disturbances;
2. High risk of death within 5 days per clinician assessment, or presence of treatment-limiting directives;
3. Active gastrointestinal bleeding or perforation indicating severe intestinal barrier damage;
4. Inability to tolerate enteral nutrition supplying ≥50% of caloric needs due to fibrotic bowel stenosis or high-output fistula;
5. Planned or recent abdominal surgery (within 14 days before enrollment);
6. Diagnosed fulminant colitis or toxic megacolon;
7. Neutropenia (absolute neutrophil count < 1500 cells/µL);
8. Congenital or acquired immunodeficiency;
9. Recent use of high-risk immunosuppressive or cytotoxic agents: e.g., rituximab, doxorubicin, or corticosteroids ≥20 mg/day prednisone equivalent for ≥4 weeks;
10. Pregnant or breastfeeding individuals;
11. Enrollment in another clinical trial within 3 months before or at study entry.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dynamic changes in the total SOFA score | Within 24 hours before FMT intervention, and on days 12, 3, 4, 5, 6 and 7 after FMT initiation
  Change in total SOFA score from randomization (baseline) to 168 hours post-intervention

SECONDARY OUTCOMES:
Changes in pulmonary microbiota diversity | Within 24 hours before FMT intervention, and at 24, 72, 120 and 168 hours after FMT initiation
  Metagenomics profiling of BALF was conducted to compare the pulmonary microbiota between the two groups. Metagenomic sequencing will be performed to analyze the dynamic changes in α-diversity (Shannon index), β-diversity, and the relative abundance of specific microbial taxa, including the Firmicutes-to-Bacteroidetes ratio, and potential pathogens.
Changes in intestinal microbiota diversity | Within 24 hours before FMT intervention, and at 24, 72, 120 and 168 hours after FMT initiation
  Metagenomics profiling of rectal swabs was conducted to compare the gut microbiota between the two groups. Metagenomic sequencing will be performed to analyze the dynamic changes in α-diversity (Shannon index), β-diversity, and the relative abundance of specific microbial taxa, including the Firmicutes-to-Bacteroidetes ratio, and potential pathogens.
Alterations in serum metabolites | Within 24 hours before FMT intervention, and at 24, 72, 120 and 168 hours after FMT initiation
  Serum samples were collected for metabolomics analysis to comprehensively examine the composition and changes of endogenous small molecule metabolites in the blood.
Change in the respiratory subscore of SOFA | Within 24 hours before FMT intervention, and on days 12, 3, 4, 5, 6 and 7 after FMT initiation
  Change in the respiratory subscore of SOFA from randomization (baseline) to 168 hours post-intervention
Correlation between gut microbiota and pulmonary microecology | Within 24 hours before FMT intervention, and at 24, 72, 120 and 168 hours after FMT initiation
  The results obtained from metagenomic and metabolomic analyses of rectal swabs and BALF were used to explore the relationship between the two
Serum lipopolysaccharide (LPS) | Within 24 hours before FMT intervention, and on days 1-3, 5, and 7 after inclusion
  The determination of serum LPS is used as an indicator for evaluating intestinal barrier function.
Serum diamine oxidase (DAO) | Within 24 hours before FMT intervention, and on days 1-3, 5, and 7 after inclusion
  The determination of serum DAO is used as an indicator for evaluating intestinal barrier function.
Serum D-lactic acid | Within 24 hours before FMT intervention, and on days 1-3, 5, and 7 after inclusion
  The determination of serum D-lactic acid is used as an indicator for evaluating intestinal barrier function.
Serum Citrulline | Within 24 hours before FMT intervention, and on days 1-3, 5, and 7 after inclusion
  The determination of serum Citrulline is used as an indicator for evaluating intestinal barrier function.
Changes of APACHE Ⅱ score | Within 24 hours before FMT intervention, and on days 1-7 after inclusion
  The APACHE II scoring system serves as a critical tool for evaluating the clinical status and prognosis of ICU patients. This system comprises three components: the Acute Physiology Score (APS), the Age Score, and the Chronic Health Evaluation Score. The total score is derived by summing these three components. The theoretical maximum score is 71, with higher scores indicating more severe conditions. Notably, the APS encompasses 12 physiological parameters and introduces a formula for calculating the risk of death (R). By aggregating the R values of all patients and dividing by the total number of patients, the predicted mortality rate for the patient population can be estimated.
Length of stay in the ICU | From date of randomization until the date of discharge from the ICU or date of death from any cause during ICU stay, whichever came first, assessed up to 6 weeks
  Duration of ICU treatment for the patient
ICU mortality rate | From date of randomization until the date of discharge from the ICU or date of death from any cause during ICU stay, whichever came first, assessed up to 6 weeks
  Mortality rate in ICU
In-hospital mortality rate | From date of randomization until the date of discharge from the hospital or date of death from any cause during hospitalization, whichever came first, assessed up to 6 weeks
  Mortality rate during hospitalization
28-day all-cause mortality rate | Within 28 days after inclusion
  The mortality rate within 28 days after inclusion in the study
90-day all-cause mortality rate | Within 90 days after inclusion
  The mortality rate within 90 days after inclusion in the study
90-day post-discharge readmission rate | Within 90 days after inclusion
  The proportion of patients readmitted within 90 days after discharge among those enrolled in the study
Secondary pulmonary infection rate within 90 days of study enrollment | Within 90 days after inclusion
  The incidence of secondary pulmonary infection within 90 days following study enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: No